CLINICAL TRIAL: NCT00582725
Title: Phase II Trial of Rituximab-CHOP (R-CHOP) Plus GM-CSF for Previously Untreated Diffuse Large Cell Lymphoma in the Elderly
Brief Title: R-CHOP + GM-CSF for Previously Untreated LCL in Elderly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HO02401; NCI-2011-00578 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2014-05

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
Keywords: DLBCL, Elderly; previously untreated DLBCL in the elderly
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- R-CHOP + GM-CSF (Experimental): R-CHOP therapy (6-8 cycles) with GM-CSF
  Interventions: Drug: R-CHOP+GM-CSF

INTERVENTIONS:
Drug: R-CHOP+GM-CSF — addition of GM-CSF

SUMMARY:
Patients will receive 6 to 8 cycles of R-CHOP (Rituximab, Cyclophosphamide, doxorubicin, vincristine, and prednisone), with GM-CSF.

DETAILED DESCRIPTION:
The objective of this study is to estimate complete response rates for patients treated with this regimen, to assess overall response rates, event-free survival and overall survival; and to assess toxicities associated with R-CHOP + GM-CSF. Patients will receive 6 to 8 cycles of R-CHOP (Rituximab, Cyclophosphamide, doxorubicin, vincristine, and prednisone), with GM-CSF.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, CD20+ B cell diffuse large cell lymphoma, with measurable or evaluable disease
* Having no prior chemotherapy, immunotherapy or radiotherapy except for one cycle of CHOP or R-CHOP.

Exclusion Criteria:

* Pregnant
* Hepatitis B Surface Antigen positive
* Have known CNS disease or HIV infection
* Have NY Classification III or IV disease.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2002-03; Primary Completion 2005-12 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Response Rate to Therapy | Dec 2005 approx

CONTACTS AND LOCATIONS:
Overall Officials: Brad Kahl, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University Of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- [Result] Kahl BS, Bailey HH, Smith EP, Turman N, Smith J, Werndli J, Williams EC, Longo WL, Kim KM, McGovern J, Jumonville A. Phase II study of weekly low-dose paclitaxel for relapsed and refractory non-Hodgkin's lymphoma: a Wisconsin Oncology Network Study. Cancer Invest. 2005;23(1):13-8. PMID 15779863